CLINICAL TRIAL: NCT07355179
Title: PLAY UP: An Intervention Program to Foster Physical Literacy Through Active Play and Environmental Affordances
Brief Title: PLAY UP: An Intervention Program Through Active Play and Environmental Affordances
Acronym: PLAY UP
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Évora (Other)
Responsible Party: Principal Investigator, Gabriela Almeida, PhD, University of Évora
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: #24101
Record Dates: First submitted 2025-12-29; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Children With Typical Neurodevelopment
Keywords: childhood; psychomotor intervention; motor competence; socialemotional competences; executive functions; physical activity; Physically active play
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- participant group (Experimental): Children in the experimental group will receive a 15-session intervention. Intervention will be implemented in the outdoors of the kindergarten, by a psychomotor therapist and children's educator. Sessions will involve active play and will prioritize, strengthen and expand opportunities for children to engage with their surroundings.
  Interventions: Behavioral: PLAY UP
- Comparison group (No Intervention): This group will maintain their regular school routine.

INTERVENTIONS:
Behavioral: PLAY UP — The PLAY UP intervention comprises 15 outdoor sessions (60 minutes each), delivered twice weekly by a psychomotor therapy professional, with the classroom educator providing pedagogical support. Sessions adopt a co-creation approach, actively engaging children in shaping play experiences while leveraging environmental affordances that promote movement and social interaction. Each PLAY UP session follows a structure, beginning with a warm-up that allows children to move freely and explore environmental affordances through active play. The main section combines guided reflection, child-led activity choices, and collective movement exploration, with adults facilitating engagement and expanding play possibilities. Sessions conclude with a symbolization and meaning-making phase, supporting reflection on experiences and promoting meaningful learning.
  Arms: participant group

SUMMARY:
The goal of this cluster-randomized trial is to investigate how a co-created, affordance-based approach - developed in collaboration with children - and combined with educator training, can support preschool children's engagement in active play and their holistic development.

ELIGIBILITY:
Inclusion Criteria:

* regular attendance in preschool; have no limitations to participate in intervention.

Exclusion Criteria:

* participating in a similar intervention program for at least 3 months; having limitations (e.g. physical limitations; intellectual neurodisorder) to take the assessment tasks;

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2026-02-23 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
physical literacy (motor competence) | 2 months
  Children's physical literacy will be assessed using Movement Assessment Battery for Children and interviews. Movement ABC consists of 3 subtests that measure three different areas: Manual dexterity; Aiming and grasping; and Balance. Assessed using the Movement Assessment Battery for Children (total standardized score derived from manual dexterity, aiming and grasping, and balance).
Physical literacy (affective/experiential domain) | 2 months
  Photo Elicitation Interviews will be conducted in small groups to ask children enjoyable experiences, appreciation, and connection to the environment, in relation to movement, play and physical activity.
Social-emotional competencies (parent-reported) | 2 months
  Strengths and Difficulties Questionnaire (SDQ), a 25- item psychosocial questionnaire completed by parents, assesses strengths, difficulties, and behavioral indicators of potential mental health issues. The SDQ total difficulties score will be used, with higher scores indicating greater behavioral difficulties.

SECONDARY OUTCOMES:
Social, Emotional, and Behavioral Competences (educator-reported) | 2 months
  Preschool and Kindergarten Behavior Scale (PKBS), completed by preschool educators, evaluates children's social-emotional skills and behavior problems during free play with their peers. The PKBS Social Skills total score will be used, with higher scores indicating better social-emotional competence.
Executive Functioning | 2 months
  Key executive functions inhibitory control, cognitive flexibility, and working memory will be assessed using the Head-Toes-Knees-Shoulders (HTKS) task. Task performance also relies on the child's sustained attention. A single composite score will be calculated combining inhibitory control, cognitive flexibility, and working memory. A higher score reflects a better executive functioning.
Physical Activity | 2 months
  Children's Physical Activity (PA) will be measured by accelerometry. Data collection will occur over one-week (on weekdays), during which children will wear accelerometer during the data collection recess. Data were normalized according to the daily hours/minutes of accelerometer use. The following cut-points were applied to classify PA intensity: sedentary (≤ 100 counts·min-¹), light (101 - 2240 counts·min-¹), moderate (2241 - 3840 counts·min-¹), and vigorous (≥ 3841 counts·min-¹) activity. The PA outcome will be minutes per day of moderate-to-vigorous physical activity (MVPA) derived from accelerometry. Sedentary, light, moderate, and vigorous activity categories are used for classification purposes.
Positional Interactions | 2 months
  Real-time spatial positioning will be continuously tracked over ~30min (during recess) using high-resolution sensor technology, capturing detailed movement trajectories and social positioning in the playground environment. Outcomes will include mean inter-child distance and frequency of proximity interactions during recess.

CONTACTS AND LOCATIONS:
Locations (1):
- Gabriela Almeida, Evora, Évora District, Portugal

IPD SHARING:
Plan to Share IPD: No
ongoing